CLINICAL TRIAL: NCT02847546
Title: Evaluation of the BARD® True™ Flow Valvuloplasty Perfusion Catheter for Aortic Valve Dilatation
Acronym: True™Flow
Status: Completed | Type: Observational
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Other Study IDs: BPV-14-004
Record Dates: First submitted 2016-07-18; First posted 2016-07-28 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: True™ Flow Valvuloplasty Perfusion Catheter — Balloon Aortic Valvuloplasty as preparation step in implantation of a Tanscatheter Aortic Valve Implantation (TAVI).

SUMMARY:
The primary objective of this study is to collect data to confirm the performance and safety of the True™ Flow Valvuloplasty Perfusion Catheter during dilatation of the aortic valve in the preparation for Transcatheter Aortic Valve Implantation (TAVI).

DETAILED DESCRIPTION:
The BARD® True™ Flow Valvuloplasty Perfusion Catheter Study is a prospective, single-center, non-randomized, single-arm observational study intended to collect data to confirm the performance and safety of the BARD® True™ Flow Valvuloplasty Perfusion Catheter (True™ Flow catheter) when used for dilatation of the aortic valve in preparation for Transcatheter Aortic Valve Implantation (TAVI). This study will be conducted in conformance with the Declaration of Helsinki, applicable national privacy laws, and European, national regulations and International Organization for Standardization (ISO) requirements (ISO 14155:2011 (E)).

ELIGIBILITY:
Inclusion Criteria:

* The subject voluntarily provides written informed consent prior to the collection of study-specific data or performance of study-specific procedures using an Informed Consent Form (ICF) that is reviewed and approved by the Ethics Committee (EC) for the site.
* The subject is a male or non-pregnant female ≥ 18 years old.
* The subject is undergoing TAVI for treatment of aortic stenosis.
* The subject has an annulus diameter that can be treated with the available size device, in accordance with the Instructions For Use (IFU).

Exclusion Criteria:

* The patient is unable or unwilling to provide written informed consent.
* The patient has a known allergy or sensitivity to contrast media that cannot be adequately pre-medicated.
* The patient has had previous aortic valve replacement.
* The patient has a known congenital aortic valve abnormality (e.g., bicuspid aortic valve).
* The patient has echocardiographic evidence of intracardiac mass, or thrombus.
* The patient has vascular conditions that make insertion and endovascular access to the aortic valve impossible.
* The patient has another medical condition, which, in the opinion of the Investigator, may cause him/her to confound the data interpretation, or is associated with a life expectancy insufficient to allow for the completion of study procedures.
* The subject is currently participating in an investigational drug, biologic, or another device study that has not completed the study treatment or that clinically interferes with the objectives of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be males or non-pregnant females, at least 18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2016-09; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Successful dilatation of the aortic valve using the True™ Flow Valvuloplasty Perfusion Catheter. | Duration of Dilatation of Balloon during Procedure (<120 minutes)
  Defined as complete opening of the True™ Flow Valvuloplasty Perfusion Catheter by visual estimate and the ability of the inflated True™ Flow Valvuloplasty Perfusion balloon to stay stationary with clinically acceptable intraventricular pressure under rapid pacing, reduced pacing, or without pacing.
Freedom from device-related or procedure-related death, stroke, annulus rupture, coronary occlusion, ventricular perforation, during the pre-dilatation procedure. | Duration of Dilatation of Balloon during Procedure (<120 minutes)
  Defined as the time the study device catheter is introduced until the time TAVI device system is introduced.

CONTACTS AND LOCATIONS:
Overall Officials: Axel Linke, Prof.Dr.med., Principal Investigator — Helios Health Institute GmbH
Locations (1):
- Leipzig Heart Institute GmbH, Leipzig, Germany

IPD SHARING:
Plan to Share IPD: Undecided